CLINICAL TRIAL: NCT00415870
Title: Ecological Momentary Intervention of Diet Via Mobile Technology
Brief Title: mDiet - Ecological Momentary Intervention of Diet Via Mobile Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kevin Patrick, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21CA115615-01A1 (NIH); 2005-4148 UCSD Number
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Overweight
Keywords: Overweight; Cell Phone; Technology
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PACE (Experimental): Received text messages and counseling calls
  Interventions: Behavioral: Printed Material; Behavioral: Weekly Weighing; Behavioral: Cell phone will serve as a self monitoring device; Device: Text Message; Behavioral: Diet Goals via Cell Phone; Behavioral: Food Monitoring
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Printed Material — Printed Material
  Arms: PACE
Behavioral: Weekly Weighing — Weekly Weighing
  Arms: PACE
Behavioral: Cell phone will serve as a self monitoring device — Cell phone will serve as a self monitoring device
  Arms: PACE
Device: Text Message — Text Message
  Arms: PACE
Behavioral: Diet Goals via Cell Phone — Diet Goals via Cell Phone
  Arms: PACE
Behavioral: Food Monitoring — Food Monitoring
  Arms: PACE

SUMMARY:
This is a NCI funded study which will develop and evaluate a cell phone application (mDIET) that can be used as an assessment and intervention tool to improve dietary behaviors and thus reduce weight in overweight and moderately obese (BMI 25-34.9) men and women ages 25-55.

DETAILED DESCRIPTION:
This research will develop a technologically advanced system for monitoring and intervening on diet behaviors (e.g., food intake, weight). Interventions aimed at dietary change are missing a comparable, portable tool. Mobile technologies can help fill this gap by providing portable connectivity to expert systems that create specific tailored diet goals based on participant profiles. The expert system can 'push' intervention messages throughout the day during critical point-of-decision moments to aid in decision making among users. The portable device can 'pull' information through prompts and easy-to-use recording. This ecological momentary assessment + ecological momentary intervention format may further encourage healthy behaviors by prompting at critical decision points to improve dietary behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they:

  * Are age 25-55
  * Are overweight or moderately obese
  * Are with a BMI between 25.0-34.9 (as defined by the NIH report on Obesity (NIH 1998)
  * Are able to read (completion of at least the 6th grade) and speak English
  * Provide consent
  * Do not intend to become pregnant or move out of the county for the duration of the intervention (16 weeks).
* Participants will also be required to have a cell phone that is capable of supporting the mDIET application.
* Participants may be otherwise healthy or have one or more risk factors for CVD, including uncomplicated Type 2 diabetes but will not be enrolled if they have diagnosed CVD.

Exclusion Criteria:

Participants will be excluded from the study if they have any of the following conditions:

* An eating disorder
* Are currently pregnant
* Have a strict dietary regimen prescribed by their doctor that will not allow them to comply with intervention guidelines related to dietary changes.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Patrick, MD, MS, Principal Investigator — UCSD
Locations (1):
- UCSD Professional Suites, La Jolla, California, United States

REFERENCES:
- [Derived] Norman GJ, Kolodziejczyk JK, Adams MA, Patrick K, Marshall SJ. Fruit and vegetable intake and eating behaviors mediate the effect of a randomized text-message based weight loss program. Prev Med. 2013 Jan;56(1):3-7. doi: 10.1016/j.ypmed.2012.10.012. Epub 2012 Oct 22. PMID 23085329
- [Derived] Patrick K, Raab F, Adams MA, Dillon L, Zabinski M, Rock CL, Griswold WG, Norman GJ. A text message-based intervention for weight loss: randomized controlled trial. J Med Internet Res. 2009 Jan 13;11(1):e1. doi: 10.2196/jmir.1100. PMID 19141433

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Enhanced Usual Care
- PACE: Received text messages and counseling calls
  Food Monitoring : Food Monitoring
  Text Message : Text Message
  Cell phone will serve as a self monitoring device : Cell phone will serve as a self monitoring device
  Diet Goals via Cell Phone : Diet Goals via Cell Phone
  Weekly Weighing : Weekly Weighing
  Printed Material : Printed Material
Period: Overall Study
Arm/Group | Control | PACE
Started | 32 | 33
Completed | 26 | 26
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Control: Enhanced Usual Care: Enhanced usual care
- PACE: Intervention - SMS Messages and Lifestyle Counseling: Received text messages and counseling calls
- Total: Total of all reporting groups
Arm/Group | Control: Enhanced Usual Care | PACE: Intervention - SMS Messages and Lifestyle Counseling | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 33 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (7.5) | 47.4 (7.1) | 44.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Mean Weight (kg)
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Control:Enhanced Usual Care: Enhanced Usual Care
- PACE: Intervention - SMS Messages: Received text messages and counseling calls
Arm/Group | Control:Enhanced Usual Care | PACE: Intervention - SMS Messages
Number analyzed (Participants) | 32 | 33
kg | 87.85 (14.11) | 85.17 (18.16)

2. Secondary Outcome: Program Satisfaction
Description: Participants reported a 2 if they liked the program, 1 if they felt neutral about the program, and 0 if they did not like program. Higher scores reflect greater satisfaction.
Time Frame: 4 months
Population: Participants in the control condition did not receive the program satisfaction survey. For those in the PACE-intervention arm, it was not mandatory to complete the program satisfaction survey and thus the number of participants who completed it are reflected in the data submitted.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control:Enhanced Usual Care | PACE: Intervention - SMS Messages
Number analyzed (Participants) | 0 | 24
score on a scale |  | 1.88 (.44)

3. Secondary Outcome: Compliance With Food Monitoring Activities
Time Frame: 4 months
Population: We did not collect these data from the phone nor reported them in our main outcome paper. To the best of our recollection we shifted our emphasis from recording types of food and amounts of food to the behaviors of eating that were reflected in the Eating Behavior Inventory (O'Neill et al, 1979; citation #20 in the main outcome paper).
Arm/Group | Control:Enhanced Usual Care | PACE: Intervention - SMS Messages
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control | PACE
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No